CLINICAL TRIAL: NCT01210755
Title: Reversion of the Anticoagulant Effect of the New Antithrombotic Agents Anti-Xa and Anti IIa by Specific and Non-specific Haemostatic Drugs,: an Ex-Vivo Study in Healthy Volunteers
Brief Title: Study in Healthy Volunteers of the Reversion by Haemostatic Drugs of the Anticoagulant Effect of New Anti-thrombotics
Acronym: REVNEWANTICO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: F. Marie, University Hospital, Grenoble
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DCIC 10 09
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Venous Thromboembolism
Keywords: Antithrombotics; Haemostatics; Antidote
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban then Dabigatran (Experimental): Cross-over study with 15 days between administration of Rivaroxaban and Dabigatran
  Interventions: Drug: Rivaroxaban, Dabigatran
- Dabigatran then Rivaroxaban (Experimental): Cross-over study with 15 days between administration of Dabigatran and Rivaroxaban
  Interventions: Drug: Dabigatran; Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban, Dabigatran — Rivaroxaban: One dose of 20mg (2 tablets of 10mg) then Dabigatran: One dose of 150mg(2 capsules of 75mg) two weeks later
  Other Names: Xarelto; Pradaxa
  Arms: Rivaroxaban then Dabigatran
Drug: Dabigatran; Rivaroxaban — Dabigatran: One dose of 150mg(2 capsules of 75mg) then Rivaroxaban: One dose of 20mg (2 tablets of 10mg)two weeks later
  Other Names: Pradaxa; Xarelto
  Arms: Dabigatran then Rivaroxaban

SUMMARY:
The purpose of this study is to evaluate whether the effect of the two new anticoagulants, Dabigatran and Rivaroxaban, can be reversed by non-specific and specific inhibitors. For Dabigatran the investigators will test the non-specific inhibitors: prothrombin complex concentrate (PCC), recombinant activated coagulation factor VII, and activated prothrombin-complex (FEIBA). For Rivaroxaban the investigators will test a specific Rivaroxaban decoy (FXa-GLAless). This will be done in a laboratory using blood plasma from healthy male volunteers.

DETAILED DESCRIPTION:
Background and objective:

Currently the most widely prescribed long term anticoagulant drugs are anti vitamin K agents (AVK). They should be used with caution because they are drugs that have a narrow therapeutic range: the difference between the effective dose and toxic dose is small. Their use thus requires careful laboratory monitoring. They can cause bleeding complications in the case of overdose. The AVKs have two antidotes: Vitamin K and prothrombin complex concentrates (PCC). These reverse the anticoagulant effect.

In recent years, new types of anticoagulants have been marketed in particular Rivaroxaban (Xarelto ®) and Dabigatran (Pradaxa ®). The way they act is different from that of AVK. They have the advantage of having a wider therapeutic range. Their use is therefore easier. They do not require such regular monitoring. However, currently, no antidote has been evaluated to reverse the effect of these anticoagulants in case of emergency.

The purpose of this study is to evaluate whether the effect of the two new anticoagulants can be reversed by non-specific and specific inhibitors. For Dabigatran we will test the non-specific inhibitors prothrombin complex concentrate (PCC), recombinant activated coagulation factor VII, and activated prothrombin complex (FEIBA). For Rivaroxaban we will test a specific Rivaroxaban decoy (FXa-GLAless). This will be done in a laboratory using blood plasma from healthy volunteers.

Methods:

This is a proof of concept, single centre, randomized, open, controlled, cross-over,phase IV study involving 10 healthy volunteers Each volunteer will be asked to attend an enrolment visit in which they will be given information about the study and asked to sign a written consent form. They will have an electrocardiogram test, their blood pressure and pulse will be measured, their medical history noted, and samples of blood and of urine will be taken.

At the second visit they will be given one dose of either Rivaroxaban (20mg) or of Dabigatran (150mg), allocated randomly, and 5 samples of blood (in total 67.5mL)will be taken over a period of 4 hours via a catheter. The blood samples will be immediately centrifuged and frozen.

At the 3rd visit, 15 days later, the volunteer will have a medical examination prior to taking the other drug. This visit will then follow the same procedure as the 2nd visit.

At the 4th visit a medical examination will be made and blood and urine samples taken.

Plasma samples will be analysed and challenged with the inhibitors in the biochemistry and haematology departments of Grenoble University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 35 years
* Subject-free any acute or chronic disease
* Subjects who signed the written informed consent
* Subject affiliated to French social security or beneficiary of a similar health insurance scheme

Exclusion Criteria:

Any subjects with at least one of the following:

* Female
* Body mass index <19 and > 29
* Active or being treated for angina, coronary syndrome, stroke or arterial disease
* Constitutional hemorrhagic disease
* Acquired bleeding disorder
* Presenting or treated for any liver disease
* Abnormal laboratory results for liver function
* History of venous thrombotic disease
* History of heparin induced Thrombocytopenia
* Surgery in the previous month
* Surgery planned within a month
* Creatinine clearance below 60 ml / min
* Clinically significant bleeding or progressive disease at risk of increased bleeding (congenital or acquired hemorrhagic syndromes, uncontrolled severe hypertension, evolving gastrointestinal ulcerative disease, recent history of gastrointestinal ulcer, vascular retinopathy, recent intracranial or intracerebral hemorrhage, intrathecal or intracerebral vascular anomalies, brain, spinal or ophthalmological surgery recently)
* Hypersensitivity to the active substance or any excipients
* Person deprived of liberty by judicial or administrative order or person subject to an order of legal protection
* Refusal of consent

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
In vitro Reversal of anticoagulation | just before and 1, 2, 3 and 4 hours after taking medicine
  Reversal of anticoagulation by return of thrombin generation time to normal value

SECONDARY OUTCOMES:
In vitro, activated partial thromboplastin time | just before and 1, 2, 3 and 4 hours after taking medicine
  1. Thrombin time, activated partial thromboplastin time.
  2. Prothrombin time, measurement of anti Xa activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Pernod, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinical Research Centre, University Hospital Grenoble, Grenoble, France